CLINICAL TRIAL: NCT03238352
Title: A Method Development Clinical Study Investigating the Efficacy of an Experimental Oral Rinse in Providing Long Term Relief From Dentinal Hypersensitivity
Brief Title: A Study to Assess Efficacy of an Experimental Oral Rinse in Providing Long Term Relief From Dentinal Hypersensitivity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 207656
Record Dates: First submitted 2017-07-19; First posted 2017-08-03 (Actual); Results first posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Sodium Fluoride

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Test Product (Experimental): Participants will rinse twice daily (morning and evening) with 10 milliliters (mL) of oral rinse for 60 timed seconds and expectorate. No further rinsing with water will be permitted after use of the oral rinse.
  Interventions: Device: Potassium oxalate
- Negative Control (Other): Participants will rinse twice daily (morning and evening) with 10 mL of oral rinse for 60 timed seconds and expectorate. No further rinsing with water will be permitted after use of the oral rinse.
  Interventions: Drug: Sodium fluoride
- Placebo (Placebo Comparator): Participants will rinse twice daily (morning and evening) with 10 mL of oral rinse for 60 timed seconds and expectorate. No further rinsing with water will be permitted after use of the oral rinse.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Potassium oxalate — Oral rinse containing 1.5 percent (%) KOX and 0 ppm fluoride
  Arms: Test Product
Drug: Sodium fluoride — Oral rinse containing 0.02% weight by weight (w/w) sodium fluoride (NaF)
  Arms: Negative Control
Other: Placebo — Oral rinse containing 0% KOX and 0 ppm fluoride
  Arms: Placebo

SUMMARY:
To investigate the efficacy of an experimental oral rinse, containing 1.5% potassium oxalate (KOX) and 0 parts per million (ppm) fluoride in relieving dentine hypersensitivity (DH) after 8 weeks use compared with a placebo oral rinse and a commercialized fluoride oral rinse.

DETAILED DESCRIPTION:
This will be a single centre, eight week, randomized, examiner-blind, three treatment, parallel group, stratified study. It will be conducted in healthy participants, with at least two sensitive teeth that meet all of the study criteria at the Screening and Baseline visits. DH will be assessed at Baseline, and after 4 and 8 weeks twice daily treatment.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Good general and mental health with, in the opinion of the investigator or medically qualified designee: a) No clinically significant and relevant abnormalities in medical history or oral Examination and b) Absence of any condition that would impact on the participant's safety or wellbeing or affect the individual's ability to understand and follow study procedures and requirements.
* Dental Health at Screening: a) Self-reported history of DH lasting more than six months but not more than 10 Years, b) Minimum of 20 natural teeth, c) Minimum of 4 accessible non-adjacent teeth (incisors, canines, premolars), preferably in different quadrants, that meet all of the following criteria: Signs of facial/cervical gingival recession and/or signs of erosion or abrasion (EAR), Tooth with MGI score =0 adjacent to the test area (exposed dentine) only and a clinical mobility of ≤1 and tooth with signs of sensitivity measured by qualifying evaporative air assessment (Schiff sensitivity score ≥ 2).
* Dental Health at Baseline: Minimum of two, non-adjacent accessible teeth (incisors, canines, premolars), that meet all of the following criteria: Tooth with signs of sensitivity, measured by qualifying tactile stimulus (Yeaple ≤20g) and evaporative air assessment (Schiff sensitivity score ≥ 2.
* Females of childbearing potential who are, in the opinion of the investigator, practicing a reliable method of contraception. Adequate contraception is defined as abstinence, oral contraceptive, either combined or progestogen alone or injectable progestogen or implants of levonorgestrel or estrogenic vaginal ring or percutaneous contraceptive patches or intrauterine device or intrauterine system or double barrier method (condom or occlusive cap [diaphragm or cervical vault caps] plus spermicidal agent [foam, gel, film, cream, suppository]) or male partner sterilization prior to the female participant's entry into the study, and this male is the sole partner for that participant).
* Participant will be current and regular (twice daily), users of an over the counter (OTC) Monograph or cosmetic oral rinse.
* Participant will be cell phone owners so that they can contactable by SMS.

Exclusion Criteria:

* A woman who is known to be pregnant or who is intending to become pregnant over the duration of the study.
* A woman who is breast-feeding.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit or previous participation in this study.
* Recent history (within the last year) of alcohol or other substance abuse.
* An employee of the sponsor or the study site or members of their immediate family.
* Presence of chronic debilitating disease which, in the opinion of the investigator, could affect study outcomes.
* Any condition which, in the opinion of the investigator, causes xerostomia.
* Dental prophylaxis within 4 weeks of Screening.
* Tongue or lip piercing.
* Desensitizing treatment within 8 weeks of Screening (professional sensitivity, treatments and non-dentifrice sensitivity treatments).
* Gross periodontal disease, treatment of periodontal disease (including surgery) within 12 months of Screening, scaling or root planning within 3 months of Screening.
* Teeth bleaching and any teeth whitening procedures within 8 weeks of Screening.
* Tooth with evidence of current or recent caries, or reported treatment of decay within 12 months of Screening.
* Tooth with exposed dentine but with deep, defective or facial restorations, teeth used as abutments for fixed or removable partial dentures, dental implants, teeth with full crowns or veneers, orthodontic bands or cracked enamel. Sensitive teeth with contributing aetiologies other than erosion, abrasion or recession of exposed dentine.
* Sensitive tooth not expected to respond to treatment with an over-the-counter dentifrice in the opinion of the investigator.
* Use of an oral care product indicated for the relief of dentine hypersensitivity within 8 weeks of screening (Participants will be required to bring their current oral care products to the site in order to verify the absence of known anti-sensitivity ingredients).
* Daily doses of medication/treatments which, in the opinion of the investigator, could interfere with the perception of pain. Examples of such medications include analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilisers, anti-depressants, mood-altering and anti-inflammatory drugs.
* Currently taking antibiotics or has taken antibiotics within two weeks of Baseline.
* Daily dose of a medication which, in the opinion of the investigator, is causing xerostomia.
* Presence of kidney disease, hyperoxaluria, or any other condition that may be exacerbated by oxalic acid or oxalate salts.
* Presence of chronic debilitating disease which, in the opinion of the investigator, could affect study outcomes.
* Any participant who, in the judgment of the investigator, should not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2017-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Fort Wayne, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one center in USA.
Pre-assignment Details: A total of 123 participates were screened, out of which 89 participants were enrolled and randomized in the study. 34 participants were not randomized as all the 34 participants did not meet study criteria.
Groups:
- Test Product (1.5% KOX, 0 Ppm Fluoride, pH 7): Participants rinsed twice daily (morning and evening) with 10 milliliters (mL) of oral rinse (1.5% KOX, 0 parts per million [ppm] fluoride, pH 7) for 60 seconds using standard fluoride dentifrice and then expectorated. No further rinsing with water was allowed after use of the oral rinse. This regimen was performed twice daily for 8 weeks.
- Negative Control (0.02% w/w Sodium Fluoride): Participants rinsed twice daily (morning and evening) with 10 mL of oral rinse (0.02% weight by weight [w/w] sodium fluoride) for 60 seconds using standard fluoride dentifrice and then expectorated. No further rinsing with water was allowed after use of the oral rinse. This regimen was performed twice daily for 8 weeks.
- Placebo (0% KOX, 0 Ppm Fluoride, pH 7): Participants rinsed twice daily (morning and evening) with 10 mL of oral rinse (0% KOX, 0 ppm fluoride, pH 7) for 60 seconds using standard fluoride dentifrice and then expectorated. No further rinsing with water was allowed after use of the oral rinse. This regimen was performed twice daily for 8 weeks.
Period: Overall Study
Arm/Group | Test Product (1.5% KOX, 0 Ppm Fluoride, pH 7) | Negative Control (0.02% w/w Sodium Fluoride) | Placebo (0% KOX, 0 Ppm Fluoride, pH 7)
Started | 43 | 23 | 23
Completed | 43 | 20 | 22
Not Completed | 0 | 3 | 1
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population comprised of all randomized participants who received at least 1 dose of study treatment. This population was based on the treatment the participant actually received.
Groups:
- Test Product (1.5% KOX, 0 Ppm Fluoride, pH 7): Participants rinsed twice daily (morning and evening) with 10 mL of oral rinse (1.5% KOX, 0 ppm fluoride, pH 7) for 60 seconds using standard fluoride dentifrice and then expectorated. No further rinsing with water was allowed after use of the oral rinse. This regimen was performed twice daily for 8 weeks.
- Negative Control (0.02% w/w Sodium Fluoride): Participants rinsed twice daily (morning and evening) with 10 mL of oral rinse (0.02% w/w sodium fluoride) for 60 seconds using standard fluoride dentifrice and then expectorated. No further rinsing with water was allowed after use of the oral rinse. This regimen was performed twice daily for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Test Product (1.5% KOX, 0 Ppm Fluoride, pH 7) | Negative Control (0.02% w/w Sodium Fluoride) | Placebo (0% KOX, 0 Ppm Fluoride, pH 7) | Total
Number analyzed (Participants) | 43 | 23 | 23 | 89
Age, Customized [Mean (Standard Deviation); unit: Years] | 46.0 (9.27) | 41.5 (9.76) | 43.0 (8.75) | 44.1 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 19 | 23 | 79
  Male | 6 | 4 | 0 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 3
  Not Hispanic or Latino | 41 | 23 | 22 | 86
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 2 | 3 | 11
  White | 37 | 20 | 20 | 77
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Schiff Sensitivity Score
Description: The examiner assessed the participant's response to an evaporative air stimulus for each tooth using the Schiff Sensitivity Scale which was scored as follows - 0: Participant did not respond to air stimulation; 1: Participant responded to air stimulus but does not request discontinuation of stimulus; 2: Participant responded to air stimulus and requested discontinuation or moves from stimulus; 3: Participant responded to stimulus, considered stimulus to be painful, and requested discontinuation of the stimulus. A reduction in Schiff Sensitivity score will be indicative of an improvement in sensitivity.
Time Frame: Week 8
Population: The Intent-to-Treat (ITT) (N=85) population comprised of all randomized participants who received at least 1 dose of study treatment and had at least 1 post-baseline efficacy evaluation. This population was based on the treatment to which the participant was randomized.
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Test Product (1.5% KOX, 0 Ppm Fluoride, pH 7) | Negative Control (0.02% w/w Sodium Fluoride) | Placebo (0% KOX, 0 Ppm Fluoride, pH 7)
Number analyzed (Participants) | 43 | 20 | 22
Score on Scale
  Schiff score at baseline | 2.59 (0.382) | 2.68 (0.406) | 2.52 (0.361)
  Change from baseline in Schiff score at Week 8 | -1.94 (0.773) | -0.75 (0.866) | -0.64 (0.848)
Statistical Analysis 1: Comparison: Test Product (1.5% KOX, 0 Ppm Fluoride, pH 7) vs Negative Control (0.02% w/w Sodium Fluoride); Test Product versus Negative Control at Week 8 is a primary endpoint comparison; Test type: Other; p < 0.0001, ANCOVA; From ANCOVA model with treatment as factor and baseline Schiff score as covariate; Difference of Least Square mean = -1.22, 95% CI 2-sided [-1.657 to -0.782], Standard Error of Mean 0.220 — Difference is first named treatment minus second named treatment such that a negative difference favors the first named treatment
Statistical Analysis 2: Comparison: Test Product (1.5% KOX, 0 Ppm Fluoride, pH 7) vs Placebo (0% KOX, 0 Ppm Fluoride, pH 7); Test type: Other; p < .0001, ANCOVA; From ANCOVA model with treatment as factor and baseline Schiff score as covariate; Difference of Least Square mean = -1.28, 95% CI 2-sided [-1.705 to -0.858], Standard Error of Mean 0.213 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Test Product (1.5% KOX, 0 Ppm Fluoride, pH 7) vs Negative Control (0.02% w/w Sodium Fluoride) vs Placebo (0% KOX, 0 Ppm Fluoride, pH 7); Test Product versus Combined Control (Placebo and Negative Control) group was obtained by using estimates statement in the ANCOVA model; Test type: Other; p < 0.0001, ANCOVA; From ANCOVA model with treatment as factor and baseline Schiff score as covariate; Difference of Least Square mean = -1.25, 95% CI 2-sided [-1.600 to -0.901], Standard Error of Mean 0.176 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Tactile Threshold
Description: The examiner assessed the response to tactile sensitivity using a Yeaple probe which allowed the application of a known force to the dentin surface, starting at 10 grams (g) and rising in increments of 10g until the tactile threshold or maximum force was reached. The tactile threshold for each tooth was determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gave two consecutive 'yes' responses was recorded as the tactile threshold. The higher the tactile threshold, the less sensitive the tooth. At baseline, the maximum force used was 20g; at all subsequent visits, it was 80g.
Time Frame: Week 8
Population: The ITT (N=85) population included all participants who were randomized received at least one dose of investigational product and had at least one post-baseline efficacy evaluation. This population was based on the treatment to which the participant was randomized.
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Test Product (1.5% KOX, 0 Ppm Fluoride, pH 7) | Negative Control (0.02% w/w Sodium Fluoride) | Placebo (0% KOX, 0 Ppm Fluoride, pH 7)
Number analyzed (Participants) | 43 | 20 | 22
Grams
  Tactile threshold at baseline | 10.35 (1.289) | 10.25 (1.118) | 10.23 (1.066)
  Change from baseline at Week 8 | 61.28 (22.095) | 23.75 (35.499) | 11.59 (26.788)
Statistical Analysis 1: Comparison: Test Product (1.5% KOX, 0 Ppm Fluoride, pH 7) vs Negative Control (0.02% w/w Sodium Fluoride); Test type: Other; p < 0.0004, ANCOVA — P-value from Van Elteren test; From ANCOVA model with treatment and baseline Schiff stratification as factors and baseline tactile threshold as a covariate; Diference of Least Square mean = 37.46, 95% CI 2-sided [22.916 to 51.995], Standard Error of Mean 7.306 — Difference is the first named treatment minus second named treatment such that a positive difference favors the first named treatment
Statistical Analysis 2: Comparison: Test Product (1.5% KOX, 0 Ppm Fluoride, pH 7) vs Placebo (0% KOX, 0 Ppm Fluoride, pH 7); Test type: Other; p < .0001, ANCOVA — P-value from Van Elteren test; [statistical method as in outcome 2, analysis 1]; Diference of Least Square mean = 49.88, 95% CI 2-sided [35.791 to 63.966], Standard Error of Mean 7.079 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Test Product (1.5% KOX, 0 Ppm Fluoride, pH 7) vs Negative Control (0.02% w/w Sodium Fluoride) vs Placebo (0% KOX, 0 Ppm Fluoride, pH 7); Test Product versus Combined Control (Placebo and Negative Control) group is obtained by using estimates statement in the ANCOVA model; Test type: Other; p < .0001, ANCOVA — P-value from Van Elteren test; [statistical method as in outcome 2, analysis 1]; Diference of Least Square mean = 43.67, 95% CI 2-sided [32.001 to 55.334], Standard Error of Mean 5.862 — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- Test Product (1.5% KOX, 0 Ppm Fluoride, pH 7): Participants rinsed twice daily (morning and evening) with 10 mL of oral rinse (1.5% KOX, 0 ppm] fluoride, pH 7) for 60 seconds using standard fluoride dentifrice and then expectorated. No further rinsing with water was allowed after use of the oral rinse. This regimen was performed twice daily for 8 weeks.
Arm/Group | Test Product (1.5% KOX, 0 Ppm Fluoride, pH 7) | Negative Control (0.02% w/w Sodium Fluoride) | Placebo (0% KOX, 0 Ppm Fluoride, pH 7)
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 4/43 | 0/23 | 2/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product (1.5% KOX, 0 Ppm Fluoride, pH 7) (N=43) | Negative Control (0.02% w/w Sodium Fluoride) (N=23) | Placebo (0% KOX, 0 Ppm Fluoride, pH 7) (N=23)
LIP ULCERATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
MOUTH ULCERATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ORAL DISCOMFORT (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ORAL MUCOSAL EXFOLIATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
TRAUMATIC ULCER (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-05-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT03238352/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/52/NCT03238352/SAP_001.pdf